CLINICAL TRIAL: NCT05581849
Title: Prolonged Nightly Fasting in Individuals With Fibromyalgia: A Pilot Study
Brief Title: Prolonged Nightly Fasting in Fibromyalgia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued due to unexpected funding constraints and resource limitations.
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016726
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia
Keywords: intermittent fasting; chronic pain; quantitative sensory testing; sleep
MeSH Terms: conditions — Fibromyalgia; Intermittent Fasting; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Nightly Fasting (PNF) (Experimental): Participants will engage in the PNF (14+ hours a night of fasting and no calorie containing food or beverages) for 8 weeks.
  Interventions: Behavioral: Prolonged Nightly Fasting
- Health Education Control (HEC) (Active Comparator): Participants in HEC group will receive weekly 15-minute videos (once weekly) focused on non-diet/non-fasting health educational content for 8 weeks.
  Interventions: Behavioral: Health Education Control

INTERVENTIONS:
Behavioral: Prolonged Nightly Fasting — Participants will engage in 14+ hours a night of fasting and no calorie containing food or beverages for 8 weeks. Participants will be allotted one "cheat day" per week, during which they will not need to fast (or track their times)- the day may change weekly and will be based on participant preference. Study staff and study participants will engage in a weekly coaching call (via phone; 5-10 minutes). Weekly coaching calls will last through the duration of the 8-week intervention.
  Other Names: Intermittent Fasting
  Arms: Prolonged Nightly Fasting (PNF)
Behavioral: Health Education Control — Participants in this group will receive weekly 15-minute videos (once weekly) focused on non-diet/non-fasting health educational content for 8 weeks. Participants will be asked to review the video at their convenience, prior to their weekly coaching call (5-10 minutes) with the study staff. Weekly topics will be as follows: Week 1: Sleep hygiene, Week 2: Sun safety, Week 3: Home safety, Week 4: Driving safety, Week 5: Hydration, Week 6: Dental health, Week 7: Working environment, Week 8: Communication.
  Arms: Health Education Control (HEC)

SUMMARY:
The present randomized-controlled pilot trial will test the feasibility, acceptability, and preliminary efficacy of an 8-week prolonged nightly fasting (PNF) intervention protocol in 20 adults with fibromyalgia.

Aim 1: Evaluate feasibility and acceptability of the PNF intervention among participants with fibromyalgia.

Aim 2: Evaluate preliminary efficacy of PNF on pain severity and sensitivity, mood, sleep and inflammation.

DETAILED DESCRIPTION:
Fibromyalgia is characterized by chronic widespread pain, sleep disturbance, fatigue, negative mood, and cognitive dysfunction. It is estimated about 4 million individuals in the U.S. are affected by fibromyalgia, which results in high disability, lost productivity, and poor quality of life. Various medications have been tested, but findings suggest only small therapeutic effects with high side effects. First line evidence-based psychosocial interventions, such as cognitive behavioral therapy, also yield only small to moderate treatment effects and they require specialized personnel. Thus, there is a dire need to develop a novel approach to manage fibromyalgia symptoms with a high safety profile, are affordable, and are easily implemented by participants without extensive guidance and support from specialized personnel.

Prolonged nightly fasting (PNF) which is a type of time-restricted eating with no or minimal caloric intake for periods of time as few as 12 hours has been shown to promote various health benefits. PNF has also been demonstrated to be highly acceptable and adherable for adults with various clinical condition. Although some dietary patterns have been explored for their impact on pain, the effects of PNF on pain-related outcomes (e.g., pain severity, pain sensitivity), mood, sleep, and inflammation among individuals with fibromyalgia have not been examined. The present randomized-controlled pilot trial will test the feasibility, acceptability, and preliminary efficacy of an 8-week PNF intervention protocol in 20 adults with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* female
* able to speak, write, and read English
* classified as having fibromyalgia based upon criteria established by the most up-to-date 2016 American College of Rheumatology (ACR) Criteria for Fibromyalgia
* has a smartphone.

Exclusion Criteria:

* history of eating disorders assessed by MINI Neuropsychiatric Interview
* self-report of chronic malignant pain (e.g., cancer, HIV) or systemic inflammatory disease (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus)
* current use of melatonin or an immunosuppressant medication (e.g., steroids)
* currently pregnant, trying to get pregnant, or breastfeeding
* plans to relocate within the next 6 months
* has diabetes mellitus
* currently trying to lose weight
* currently routinely fasting more than 12 hours a night
* works night shifts

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility--drop-out rate | At 8 weeks post-treatment
Feasibility--adherence to intervention | At 8 weeks post-treatment
  The number of days prolonged nightly fasting was completed divided by the total number of treatment days
Acceptability of the intervention | At 8 weeks post-treatment
  It will be measured by the Global Satisfaction subscale in an adapted version of the Treatment Satisfaction Questionnaire for Medication. The scores are calculated for each of the subscales, which range from 0 to 100, with higher scores indicating higher patient satisfaction with the intervention.

SECONDARY OUTCOMES:
Fatigue | Baseline and 8 weeks post-treatment
  Total score of Fatigue Severity Scale (ranges from 9-63; higher score means greater fatigue severity)
Fibromyalgia symtpoms | Baseline and 8 weeks post-treatment
  Total score from Revised Fibromyalgia Impact Questionnaire (FIQR) (ranges from 0-100; higher score means greater fibromyalgia symptom severity)
Cognitive Functioning | Baseline and 8 weeks post-treatment
  Total score from Montreal Cognitive Assessment (MoCA) (ranges from 0-30; higher score means better cognitive functioning)
Pain Severity | Baseline and 8 weeks post-treatment
  Average of 4 items from the Brief Pain Inventory; each rated on a 0 (no pain) to 10 (pain as bad as you can imagine); ratings are made of pain right now, typical pain, worst pain, and least pain during the past week.
Central Sensitization Index | Baseline and 8 weeks post-treatment
  Index of thermal temporal summation, mechanical temporal summation, conditioned pain modulation, and aftersensations (this is standardized Z-score)
Pain Interference | Baseline and 8 weeks post-treatment
  Average of 7 items from the Brief Pain Inventory; assessing the extent to which participant experienced that pain interfered with their (1) general activity, (2) mood; (3) walking ability; (4) normal walk; (5) relations with other people, (6) sleep, and (7) enjoyment of life
Inflammatory levels | Baseline and 8 weeks post-treatment
  IL-1β, IL-6, and TNF-α and C-Reactive Protein (CRP) levels
Total Sleep Time (TST) | Baseline and 8 weeks post-treatment
  TST is defined as the total number of minutes asleep between the time a participant goes to bed at night and the time a participant gets out of bed in the morning. TST will be derived from ambulatory EEG sleep monitoring.
Depressive symptoms | Baseline and 8 weeks post-treatment
  T-score from PROMIS Emotional Distress-Depression-Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Chung Jung Mun, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No